CLINICAL TRIAL: NCT05623488
Title: Phase 1, Adaptive-design Trial of Human Chimeric Antigen Receptor Modified T Cells in Patients With Mesothelin Expressing Breast Cancer
Brief Title: CAR T Cells in Mesothelin-Expressing Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Feasibility Concerns
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC# 15122, IRB # 852205
Record Dates: First submitted 2022-11-11; First posted 2022-11-21 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Dose Level 1 (Experimental): 3.00 x 10^7 CAR T cells administered intratumoral
  Interventions: Drug: huCART-meso cells; Device: Mesothelin Expression Testing
- Dose Level -1 (Experimental): 3.00 x 10^6 CAR T cells administered intratumoral
  Interventions: Drug: huCART-meso cells; Device: Mesothelin Expression Testing

INTERVENTIONS:
Drug: huCART-meso cells — Autologous T cells lentivirally transduced with chimeric anti-mesothelin immunoreceptor M5 scFv fused to the 4-1BB and CD3ζ signaling domains
Device: Mesothelin Expression Testing — Laboratory Developed Test

SUMMARY:
Phase 1 - Safety and Proof of Concept

DETAILED DESCRIPTION:
This is a phase I study to establish the safety and feasibility of lentiviral transduced CAR T cell products in patients with mesothelin expressing breast cancer. This study will be initiated as a single cohort, however the study is designed to allow for additional disease indications and other investigational CAR T cell products to be explored as separate cohorts under this protocol in the future.

Cohort 1: Cohort 1 will evaluate the use of huCART-meso cells delivered intratumorally in patients with locally advanced unresectable or metastatic triple-negative breast cancer (TNBC) which is positive for mesothelin expression by IHC. Eligible subjects must also have an accessible lesion that can be targeted for both intratumoral injection and surgical excision/biopsy by either a surgeon or interventional radiology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with locally advanced unresectable or metastatic triple-negative breast cancer as confirmed by all of the following:

   1. ER-negative or low-ER positive (≤ 10% by IHC)
   2. PR-negative or low-PR positive (≤ 10% by IHC)
   3. HER2 negative by IHC/FISH
2. Patients with an accessible lesion that can be targeted for both intratumoral injection and surgical excision/biopsy by either a surgeon or interventional radiology.
3. Confirmed tumor mesothelin expression by ≥ 10% of malignant cells by IHC.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Adequate organ and bone marrow function defined as:

   1. Bilirubin ≤ 2.0 x ULN
   2. Serum Creatinine ≤ 1.5 x ULN
   3. ALT/AST ≤ 3 x ULN
   4. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and pulse oxygen > 92% on room air
   5. Left Ventricle Ejection Fraction (LVEF) ≥ 45% confirmed by echocardiogram
6. Male and female patients ≥ 18 years of age.
7. Provides written informed consent.
8. Subjects of reproductive potential must agree to use acceptable birth control methods

Exclusion Criteria:

1. Active invasive cancer other than the study-targeted malignancy.
2. Evidence of active hepatitis B or hepatitis C. The following would not qualify as an active infection, thus would not exclude the subject from participating:

   1. Positive HBV serology with undetectable viral load and ongoing antiviral prophylaxis for potential HBV reactivation.
   2. Positive HCV serology with quantitative PCR for plasma HCV RNA below the lower limit of detection, with or without concurrent antiviral HCV treatment.
3. Patients with ongoing or active infection.
4. Active autoimmune disease requiring systemic immunosuppressive treatment equivalent to ≥ 10 mg/day of prednisone. Patients with autoimmune neurologic diseases (such as MS) will be excluded.
5. Planned concurrent treatment with systemic high dose corticosteroids. Patients may be on a stable low dose of steroids (≤ 10mg daily equivalent of prednisone). Use of inhaled or topical steroids is allowable.
6. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40).
7. Pregnant or breastfeeding women.
8. Any clinically significant pericardial effusion, Class II-IV cardiovascular disability according to the New York Heart Association Classification or other cardiovascular condition that would preclude assessment of mesothelin induced pericarditis or that may worsen as a result of toxicities expected for this study. This determination will be made by a cardiologist if cardiac issues are suspected.
9. Patients with significant lung disease as follows:

   1. Patients with radiographic evidence of greater than lobar lymphangitic pulmonary involvement, greater than lobar bronchial wall thickening suggestive of peribronchial lymphatic disease extension, and/or evidence of extensive bilateral parenchymal metastatic burden.
   2. Patients with radiographic and/or clinical evidence of active radiation pneumonitis.
   3. Patients with radiographic evidence of underlying interstitial lung disease, including evidence of unresolved drug toxicity from any agent (e.g. chemotherapy, targeted agents, amiodarone, nitrofurantoin, etc).
10. Patients with active central nervous system (CNS) involvement. Screening for this (e.g. lumbar puncture, brain MRI, etc) is not required unless the patient is symptomatic and/or radiographic findings are present.
11. Patient has prior/ongoing treatment that will not accommodate washout requirements for immune checkpoint inhibitors as described in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment-limiting toxicities (TLTs) | 90 days
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0. | 15 years

SECONDARY OUTCOMES:
Proportion of manufacturing product that do not meet the release criteria. | 60 days
Proportion of the products that meet the target dose. | 60 days
Proportion of enrolled subjects that receive study treatment. | 60 days
Proportion of eligible subjects that receive study treatment | 60 days
Proportion of subjects for which standard of care treatment is not impacted due to CAR T cell related toxicity. | 90 days
Kinetics of expansion and persistence of infused cells by flow cytometry. | 90 days
Kinetics of expansion and persistence of infused cells by quantitative PCR. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Julia Tchou, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No